CLINICAL TRIAL: NCT05342597
Title: Clinical Pharmacology Study of Oral Edaravone in Healthy Adult Subjects (Food Effect Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MT-1186-J06
Record Dates: First submitted 2022-04-19; First posted 2022-04-22 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): A single oral dose of MT-1186 with fasted condition in period 1, meal 1 condition in period 2, meal 2 condition in period 3, meal 3 condition in period 4, and meal 4 condition in period 5.
  Interventions: Drug: MT-1186
- Group B (Experimental): A single oral dose of MT-1186 with meal 1 condition in period 1, meal 2 condition in period 2, meal 3 condition in period 3, fasted condition in period 4, and meal 4 condition in period 5.
  Interventions: Drug: MT-1186
- Group C (Experimental): A single oral dose of MT-1186 with meal 2 condition in period 1, meal 3 condition in period 2, fasted condition in period 3, meal 1 condition in period 4, and meal 4 condition in period 5.
  Interventions: Drug: MT-1186
- Group D (Experimental): A single oral dose of MT-1186 with meal 3 condition in period 1, fasted condition in period 2, meal 1 condition in period 3, meal 2 in period 4, and meal 4 condition in period 5.
  Interventions: Drug: MT-1186

INTERVENTIONS:
Drug: MT-1186 — A crossover study in which Japanese healthy subjects receive a single dose of MT-1186 under several dosing condition on Day 1, 3, 5, 7 and 24 according to their treatment sequence.
  Other Names: Edaravone

SUMMARY:
To evaluate the effect of food on the pharmacokinetics of oral edaravone in healthy adult subjects. In this study, we determined 5 different dietary conditions including 4 different meal contents and fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria and who have the capability of giving informed consent will be included in the study.

  1. Healthy adult male or female volunteers
  2. Japanese
  3. Subjects aged between 20 and 45 years at the time of informed consent
  4. Subjects who have thoroughly understood the contents of the study and voluntarily provided written informed consent to participate in the study

Exclusion Criteria:

* Subjects who met any of the following exclusion criteria between screening and investigational product administration were excluded from the study:

  1. Subjects with a current or previous history of cardiac, hepatic, renal, gastrointestinal, respiratory, psychiatric/nervous, hematopoietic, or endocrine diseases, and those whom the investigator (or subinvestigator) deems unsuitable for the study
  2. History of drug or food allergies
  3. History of alcohol or drug abuse or dependence
  4. Body mass index (BMI) of < 18.0 or > 30.0, or a body weight of < 50 kg [BMI formula: body weight (kg)/height (m)2, rounded to one decimal place]
  5. Positive test for any of the following at screening: hepatitis B surface (HBs) antigen, serological test for syphilis, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen/antibody
  6. Any clinically significant 12-lead ECG abnormality or corrected QT interval (QTc) using Fridericia's formula (QTcF) interval ≥ 450 msec
  7. Blood donation or sampling with a total volume of ≥ 400 mL within 12 weeks, ≥ 200 mL within 4 weeks, or ≥ 800 mL within one year before providing informed consent
  8. Blood component donation or blood sampling within 2 weeks before providing informed consent
  9. Subjects who have undergone any surgery known to affect the gastrointestinal absorption of drugs (except for appendectomy and herniotomy)
  10. Female subjects who do not agree to use an effective method of contraception from screening or 2 weeks before the start of investigational product administration, whichever comes earlier, to 14 days after the completion (or discontinuation) of investigational product administration. Male subjects who do not agree to use an effective method of contraception from the start of investigational product administration to 14 days after the completion (or discontinuation) of investigational product administration
  11. Subjects who have previously received edaravone
  12. Subjects who have participated in another clinical study and received an investigational product within 12 weeks before providing informed consent
  13. Subjects who have used any drugs other than the single use of acetylsalicylic acid within 7 days before the initiation of investigational product administration
  14. Use of any nutritional supplement(s) within 7 days before the initiation of investigational product administration
  15. Use of alcohol or any products containing xanthin or caffeine within 24 hours before screening and visit on Day -1
  16. Use of grapefruit, grapefruit juice, or any processed food(s) containing these substances within 24 hours before screening and visit on Day -1
  17. Use of any tobacco or nicotine-containing product(s) within 24 hours before screening and visit on Day -1
  18. Female subjects who have a positive pregnancy test at screening and on Day -1, are pregnant or breast feeding, or plan to get pregnant during the study
  19. Subjects judged by the investigator (or subinvestigator) to be unsuitable for the study for any other reason

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shimizu H, Nishimura Y, Shiide Y, Akimoto M, Matsuda H, Kato Y, Hirai M. Food Effect Study to Assess the Impact on Edaravone Pharmacokinetic Profiles in Healthy Participants. Clin Ther. 2022 Dec;44(12):1552-1565. doi: 10.1016/j.clinthera.2022.10.001. Epub 2022 Nov 12. PMID 36376130

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: A crossover study in which Japanese healthy subjects receive a single dose of MT-1186 under several dosing condition on Day 1, 3, 5, 7 and 24 according to their treatment sequence.
  MT-1186 orally dosing under fasted condition in period 1, dosing 8 hours after high-fat meal in period 2, dosing 4 hours after low-fat meal in period 3, dosing 2 hours after light meal in period 4, and dosing 2 hours after low-fat meal in period 5.
- Group B: A crossover study in which Japanese healthy subjects receive a single dose of MT-1186 under several dosing condition on Day 1, 3, 5, 7 and 24 according to their treatment sequence.
  MT-1186 orally dosing 8 hours after high-fat meal in period 1, dosing 4 hours after low-fat meal in period 2, dosing 2 hours after light meal in period 3, dosing under fasted condition in period 4 and dosing 2 hours after low-fat meal in period 5.
- Group C: A crossover study in which Japanese healthy subjects receive a single dose of MT-1186 under several dosing condition on Day 1, 3, 5, 7 and 24 according to their treatment sequence.
  MT-1186 orally dosing 4 hours after low-fat meal in period 1, dosing 2 hours after light meal in period 2, dosing under fasted condition in period 3, dosing 8 hours after high-fat meal in period 4 and dosing 2 hours after low-fat meal in period 5.
- Group D: A crossover study in which Japanese healthy subjects receive a single dose of MT-1186 under several dosing condition on Day 1, 3, 5, 7 and 24 according to their treatment sequence.
  MT-1186 orally dosing 2 hours after light meal in period 1, dosing under fasted condition in period 2, dosing 8 hours after high-fat meal in period 3, dosing 4 hours after low-fat meal in period 4 and dosing 2 hours after low-fat meal in period 5.
Period: Period 1
Arm/Group | Group A | Group B | Group C | Group D
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Group A | Group B | Group C | Group D
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Group A | Group B | Group C | Group D
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Group A | Group B | Group C | Group D
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Group A | Group B | Group C | Group D
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 16
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 3 | 3 | 3 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 4 | 4 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve From Zero up to Infinity (AUC0-inf) of Edaravone
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: Four groups of randomized participants received edaravone oral suspension under 5 dosing conditions (4 subjects per group, 16 subjects per dosing condition).
Measure: Mean (Standard Deviation); unit: ng·h/mL
Groups:
- Edaravone Single Dose Under Fasting Condition; Edaravone Single Dose 8 Hours After a High-fat Meal; Edaravone Single Dose 4 Hours After a Low-fat Meal; Edaravone Single Dose 2 Hours After a Light Meal; Edaravone Single Dose 2 Hours After a Low-fat Meal: Subjects receive the edaravone oral suspension orally.
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng·h/mL | 2165 (673) | 2209 (658) | 2073 (641) | 1955 (523) | 1717 (463)
Statistical Analysis 1: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 8 Hours After a High-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — Estimated difference in least squares means and corresponding 90%CI of log-transformed PK parameters were back transformed to obtain the estimate and CI of the geometric mean ratio of each meal condition to the fasted state; ANOVA; LS Mean Ratio = 1.025, 90% CI 2-sided [0.931 to 1.128]
Statistical Analysis 2: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 4 Hours After a Low-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Ratio = 0.959, 90% CI 2-sided [0.871 to 1.056]
Statistical Analysis 3: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 2 Hours After a Light Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Ratio = 0.910, 90% CI 2-sided [0.827 to 1.002]
Statistical Analysis 4: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 2 Hours After a Low-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Ratio = 0.801, 90% CI 2-sided [0.712 to 0.901]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Edaravone
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng/mL | 2318 (1229) | 2525 (1337) | 2020 (1114) | 1898 (865.9) | 1276 (805.6)
Statistical Analysis 1: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 8 Hours After a High-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Ratio = 1.083, 90% CI 2-sided [0.821 to 1.429]
Statistical Analysis 2: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 4 Hours After a Low-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Ratio = 0.872, 90% CI 2-sided [0.661 to 1.150]
Statistical Analysis 3: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 2 Hours After a Light Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Ratio = 0.820, 90% CI 2-sided [0.621 to 1.082]
Statistical Analysis 4: Comparison: Edaravone Single Dose Under Fasting Condition vs Edaravone Single Dose 2 Hours After a Low-fat Meal; PK parameters of unchanged edaravone were analyzed for the assessments of food effect on PK; Test type: Other — [test comment as in outcome 1, analysis 1]; ANOVA; LS Mean Ratio = 0.536, 90% CI 2-sided [0.362 to 0.794]

3. Primary Outcome: AUC0-inf of Sulfate Conjugate and Glucuronide Conjugate
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng·h/mL
  Sulfate conjugate | 24519 (7243) | 25724 (7729) | 24671 (6077) | 25903 (8657) | 26293 (10355)
  Glucuronide conjugate | 4054 (791) | 3895 (796) | 4109 (891) | 3914 (841) | 4325 (1054)

4. Primary Outcome: Cmax of Sulfate Conjugate and Glucuronide Conjugate
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng/mL
  Sulfate conjugate | 8456 (2041) | 9024 (2430) | 8629 (1960) | 8665 (2362) | 7986 (2288)
  Glucuronide conjugate | 2283 (496.2) | 2209 (645.9) | 2283 (486.7) | 2141 (548.1) | 2031 (608.9)

5. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Unchanged Edaravone, Sulfate Conjugate and Glucuronide Conjugate
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
h
  Unchanged edaravone | 0.38 [0.25 to 0.50] | 0.25 [0.08 to 0.75] | 0.50 [0.25 to 0.75] | 0.38 [0.25 to 1.00] | 0.50 [0.25 to 1.50]
  Sulfate conjugate | 0.75 [0.50 to 0.75] | 0.63 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 0.75 [0.50 to 1.50] | 1.00 [0.75 to 1.50]
  Glucuronide conjugate | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 0.50 [0.50 to 1.50] | 0.75 [0.50 to 1.00]

6. Primary Outcome: Terminal Elimination Half-life (t1/2) of Unchanged Edaravone, Sulfate Conjugate and Glucuronide Conjugate
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
h
  Unchanged edaravone | 8.17 (2.29) | 7.38 (1.97) | 9.05 (5.07) | 7.31 (4.3) | 11.25 (8.35)
  Sulfate conjugate | 6.32 (1.85) | 7.16 (2.52) | 5.85 (1.18) | 6.25 (1.69) | 4.91 (1.02)
  Glucuronide conjugate | 4.12 (0.34) | 4.07 (0.41) | 4.12 (0.46) | 4.03 (0.7) | 3.67 (0.34)

7. Primary Outcome: Apparent Terminal Elimination Rate Constant (Kel) of Unchanged Edaravone, Sulfate Conjugate and Glucuronide Conjugate
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
1/h
  Unchanged edaravone | 0.0931 (0.0343) | 0.0999 (0.0248) | 0.1010 (0.0645) | 0.1108 (0.0330) | 0.0864 (0.0435)
  Sulfate conjugate | 0.1164 (0.0249) | 0.1062 (0.0300) | 0.1221 (0.0195) | 0.1172 (0.0246) | 0.1463 (0.0266)
  Glucuronide conjugate | 0.1690 (0.0125) | 0.1720 (0.0162) | 0.1699 (0.0173) | 0.1762 (0.0254) | 0.1905 (0.0176)

8. Primary Outcome: Mean Residence Time (MRT) of Unchanged Edaravone
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
h | 2.35 (0.52) | 2.19 (0.49) | 2.34 (0.44) | 2.32 (0.54) | 3.55 (0.87)

9. Primary Outcome: Apparent Total Clearance (CL/F) of Unchanged Edaravone
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
L/h | 53.0 (16.3) | 51.4 (14.4) | 55.1 (16.9) | 57.9 (17.6) | 65.4 (17.3)

10. Primary Outcome: Apparent Distribution Volume at Elimination Phase (Vz/F) of Unchanged Edaravone
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
L | 608 (247) | 530 (156) | 646 (239) | 585 (305) | 993 (666)

11. Primary Outcome: Apparent Distribution Volume at Steady State (Vss/F) of Unchanged Edaravone
Time Frame: Before administration, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
L | 126.4 (57.2) | 114.2 (46.7) | 128.6 (41.6) | 136.1 (59.0) | 231.4 (84.0)

12. Primary Outcome: Cumulative Urinary Excretion Amount (Ae 0-24h) of Unchanged Edaravone, Sulfate Conjugate and Glucuronide Conjugate
Time Frame: Day 1 to 9, Day 24 to 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
mg
  Unchanged edaravone | 0.819 (0.349) | 1.609 (2.630) | 0.977 (0.406) | 0.988 (0.965) | 1.302 (2.086)
  Sulfate conjugate | 13.87 (12.62) | 13.10 (12.61) | 13.13 (13.99) | 13.14 (10.96) | 8.89 (9.50)
  Glucuronide conjugate | 144.6 (19.9) | 146.8 (20.5) | 144.0 (18.4) | 153.2 (22.6) | 160.2 (44.8)

13. Primary Outcome: Urinary Excretion Ratio (Ae% 0-24h) of Unchanged Edaravone, Sulfate Conjugate and Glucuronide Conjugate
Time Frame: Day 1 to 9, Day 24 to 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of dose
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
% of dose
  Unchanged edaravone | 0.780 (0.349) | 1.533 (2.505) | 0.931 (0.386) | 0.941 (0.919) | 1.240 (1.986)
  Sulfate conjugate | 9.08 (8.27) | 8.58 (8.26) | 8.60 (9.17) | 8.61 (7.18) | 5.82 (6.22)
  Glucuronide conjugate | 68.7 (9.5) | 69.7 (9.7) | 68.4 (8.8) | 72.8 (10.7) | 76.1 (21.3)

14. Primary Outcome: Renal Clearance (CLr) of Unchanged Edaravone
Time Frame: Day 1 to 9, Day 24 to 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
L/h | 0.419 (0.271) | 0.818 (1.413) | 0.535 (0.333) | 0.545 (0.535) | 0.871 (1.582)

15. Secondary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions
Time Frame: Day 1 to Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Number of Participants with Adverse events | 0 | 0 | 1 | 0 | 0
  Number of Participants with adverse drug reactions | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 31
Description: Four groups of randomized participants received edaravone oral suspension under 5 dosing conditions (4 subjects per group, 16 subjects per dosing condition).
Arm/Group | Edaravone Single Dose Under Fasting Condition | Edaravone Single Dose 8 Hours After a High-fat Meal | Edaravone Single Dose 4 Hours After a Low-fat Meal | Edaravone Single Dose 2 Hours After a Light Meal | Edaravone Single Dose 2 Hours After a Low-fat Meal
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 1/16 | 0/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edaravone Single Dose Under Fasting Condition (N=16) | Edaravone Single Dose 8 Hours After a High-fat Meal (N=16) | Edaravone Single Dose 4 Hours After a Low-fat Meal (N=16) | Edaravone Single Dose 2 Hours After a Light Meal (N=16) | Edaravone Single Dose 2 Hours After a Low-fat Meal (N=16)
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT05342597/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT05342597/SAP_001.pdf